CLINICAL TRIAL: NCT06835699
Title: Open Label Psilocybin Brain Stimulation and Imaging Pilot Study
Brief Title: Psilocybin Brain Stimulation and Imaging Pilot Study
Acronym: OPTE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00451481
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Psilocybin and TMS (Experimental): All participants will be administered 25 mg psilocybin and undergo TMS
  Interventions: Drug: Psilocybin 25 mgs; Device: TMS

INTERVENTIONS:
Drug: Psilocybin 25 mgs — All participants will be administered 25 mg psilocybin and undergo TMS
Device: TMS — All participants will be administered 25 mg psilocybin and undergo TMS

SUMMARY:
This open-label pilot psilocybin administration study investigates the influence of psilocybin on brain function and cognitive control functions in clinically and psychiatrically healthy volunteers. Participants will undergo experimental drug administration sessions after careful screening and preparation. Participants will also have brain activity measured using electroencephalogram (EEG) also during non-invasive brain stimulation using Transcranial Magnetic Stimulation (TMS).

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Right handed
* Between the ages of 22 and 55 years old
* Have a high school level of education
* Be medically healthy and psychologically stable as determined by screening for medical problems via a personal interview, medical history and physical examination, psychiatric interview, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests
* Fluent in English and capable of providing informed consent
* Willing to remove any jewelry, hair clips, bobby pins, or any other potentially conducting or magnetic objects worn on or near the head
* Have a minimum of 2 lifetime uses of a hallucinogen (e.g., Lysergic acid diethylamide (LSD), psilocybin mushrooms, N,N-dimethyltryptamine (DMT), ayahuasca, mescaline, Salvia divinorum, ketamine, dextromethorphan (DXM) , and phencyclidine (PCP). Only psychoactive and recreational use of the hallucinogenic drugs, including dextromethorphan and ketamine, will be factored into the calculation of lifetime use.
* Cigarette smokers must agree to abstain from smoking on session days from 1 hour before drug administration
* Agree to refrain from using any psychoactive drugs, including alcoholic beverages, within 24 hours of each drug administration. Exceptions include daily use of caffeine and nicotine.
* Agree that for one week before each session, he/she will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except if approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals
* Agree not to take any "as-needed", pro re nata (PRN) prescription medications on the mornings of the sessions
* Agree not to operate dangerous machinery or a motor vehicle for at least 12 hours after leaving the research unit
* (for male participants) Agree to use contraception and refrain from sperm donation within two weeks of completing dosing sessions, as the reproductive safety for psilocybin is not yet established. Effective methods of contraception are barrier, hormonal and sterilization methods.
* (for female participants) Agree to use highly effective birth control measure within two weeks of completing the dosing sessions. Effective methods of contraception are barrier, hormonal and sterilization methods.

Exclusion Criteria:

* Weight greater than 350 lbs (the weight limit of the specialized TMS/EEG chair)
* Weight less than 40 kg
* Cardiovascular conditions: coronary artery disease, stroke, angina, hypertension with resting blood pressure systolic >139 or diastolic >89, a clinically significant ECG abnormality (e.g., atrial fibrillation), prolonged corrected QT (QTc) interval (i.e., QTc > 450 msec), artificial heart valve, or Transient Ischemic Attack (TIA) in the past year
* Hallucinogen use within the past 6 months (preference given to volunteers who have maintained a longer period of abstinence).
* Epilepsy with history of seizures
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Current or past history of meeting Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria for schizophrenia, psychotic disorder (including of substance-induced but excluding due to a medical condition), dissociative disorder, bipolar I or II disorder, or an eating disorder
* Have tinnitus or other hearing problems
* Have a first degree relative with schizophrenia, psychotic disorder (unless substance induced or due to a medical condition), or bipolar I or II disorder
* Have a first degree relative with a history seizures, epilepsy, or acute spells of unknown origin
* Have an intracranial lesion
* Have suffered ischemic or hemorrhagic stroke
* Currently taking psychoactive prescription medication on a regular (e.g., daily) basis
* Currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting pharmacological effect on serotonin neurons or medications that are monoamine Oxidase (MAO) inhibitors. For individuals who have intermittent or PRN use of such medications, sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose
* Currently taking the antiviral drug, efavirenz
* Acute intoxication with any drug of abuse, including alcohol or cannabis
* Current or past-year substance use disorder
* Pregnancy
* History of neurological problems, including epilepsy, seizures, syncope, tinnitus, migraine, or frequent non-migraine (e.g. tension) headaches
* History of head trauma associated with loss of consciousness
* Language or hearing impairment that would undermine communication regarding consent, study procedures, and overall volunteer safety.
* Irritable skin
* TMS-contraindicated medical devices, including cochlear implants, pacemaker, neurosensory stimulator, implantable defibrillator, insulin pump, clips, stents, or shunts that may be disrupted by or interact with TMS coil operation
* Taking medications that lower seizure threshold
* MRI contraindications (e.g. claustrophobia incompatible with MRI scanning, medical device or implant incompatible with MRI, prior history as a metal worker and/or certain metallic objects in the body -- must complete MRI screening form and be approved by MRI technologist before the scan

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Acute Change in Inhibitory EEG Component Amplitudes (N45, N100) from Baseline | Baseline up to approximately 1.5 hours post psilocybin adminstration
  Change in the amplitudes of inhibitory event-related potentials (ERPs), specifically the N45 and N100 components, from baseline to peak acute subjective effects (~1.5 hours post-psilocybin administration) will be calculated. This is a continuous variable expressed in microvolts (µV), derived from EEG recordings.
Change in Mystical Experience Questionnaire (MEQ30) | Baseline up to to approximately 1.5 hours post psilocybin administration
  The Mystical Experience Questionnaire was developed to assess phenomenological content during altered states of consciousness. Change in MEQ30 from baseline to peak acute psilocybin effects (~1.5 hr post-psilocybin administration) will be calculated. Score range 0 - 150 with higher scores reflecting more mystical experience.

CONTACTS AND LOCATIONS:
Overall Officials: Ceyda Sayali, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States